CLINICAL TRIAL: NCT02908360
Title: Study of the Frequency and of the Regulatory Function of Positive T Lymphocytes Dual CD4CD8aa (DP8a) Specific to a Bacteria of the Intestinal Microbiota (Faecalibacterium Prausnitzii) in Atopic Dermatitis, Asthma and Allergic Rhinitis
Acronym: Prévall-DP
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0372
Record Dates: First submitted 2016-09-09; First posted 2016-09-21 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Allergic Asthma; Allergic Rhinitis; Atopic Dermatitis
Keywords: Double positive lymphocyte T F prausnitzii
MeSH Terms: conditions — Rhinitis, Allergic; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMC
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with allergic rhinitis: Patients with rhinitis and / or allergic conjunctivitis duly diagnosed according to the ARIA criteria
  Interventions: Genetic: double positive T cells (CD4 + / CD8 +) to the specific peripheral blood of F prauznitzii analyse
- Patients with atopic dermatitis: The patient has moderate classified atopic dermatitis (SCORAD 25 to 50) or severe (SCORAD> 50).
  Interventions: Genetic: double positive T cells (CD4 + / CD8 +) to the specific peripheral blood of F prauznitzii analyse
- Patients with allergic asthma: The patient has allergic asthma diagnosed according to the criteria GINA21
  Interventions: Genetic: double positive T cells (CD4 + / CD8 +) to the specific peripheral blood of F prauznitzii analyse

INTERVENTIONS:
Genetic: double positive T cells (CD4 + / CD8 +) to the specific peripheral blood of F prauznitzii analyse

SUMMARY:
The prevalence of allergic diseases (atopic dermatitis, asthma, rhinitis, conjunctivitis and food allergy) has increased dramatically in industrialized countries over the last 20-30 years.

Allergic diseases are present especially in children and young adults, but all age groups are affected, with variations across countries and age. To propose new therapies, the investigators must first understand the physiopathology.

Since their discovery the regulatory T cells have continued to be the subject of work to understand their role in maintaining immune homeostasis in the human body but also their involvement in autoimmune diseases, inflammatory diseases, transplants of solid organs or fluids and allergic diseases.

It was identified two broad classes of regulatory T cells:

* T cells = natural regulators acquisition of a phenotype and a regulatory function right out of the thymus ( CD25 + / CD127 + low / FoxP3 +).
* T cells induced regulators = acquisition of a phenotype and a regulatory function on the periphery depending on the cytokine micro-environment.

Phenotypic characterization of these is less obvious and even more so than during the last ten years several induced regulatory T cell populations have been described ( eg, Tr1 ).

A new subpopulation of T cells induced in patients with inflammatory bowel disease recently identified have a particular phenotype as bearing the CD4 and CD8 double marking with a regulatory phenotype.

These regulatory T cells are also induced a specific of a commensal intestinal bacterium (Faecalibacterium prausnitzii).

Regarding allergies, it has been widely demonstrated a relationship between changes of the intestinal microbiota and the occurrence of allergic diseases.

The investigators would therefore propose a cross-sectional study, single-center, controlled, single blinded to study the role of T cells called double positive induced regulators DP8 to compare the frequency and the regulatory function of specific DP8 of Faecalibacterium prausnitzii in atopic dermatitis, asthma and allergic rhinitis compared to control samples.

DETAILED DESCRIPTION:
The primary endpoint will be the highlight of a quantitative reduction of double positive T cells (CD4 + / CD8 +) the specific F prausnitzii peripheral blood in patients with allergic asthma, allergic rhinitis and atopic dermatitis compared to samples from a control sample collection made available by the laboratory BIOFORTIS® located near Nantes University of Nantes.

ELIGIBILITY:
Inclusion Criteria:

* non smoker
* BMI <30kg/m²
* No contraindication to prick-test
* Inform consent signed for genetics
* belong to a social security scheme
* patients with allergic rhinitis or atopic dermatitis or with allergic asthma

Exclusion Criteria:

* major or major incapable protected
* antimicrobial treatment (antibiotic, antifungal or antiviral)
* in contact with an MDR bacteria
* has received or is receiving specific immunotherapy
* History of cancer of the hematopoietic system
* antecedent acquired immune deficiency with HIV
* congenital immunodeficiency
* inflammatory bowel disease
* autoimmune disease and / or inflammatory
* solid organ transplant or hematopoietic cells
* addict
* pregnant or of childbearing age without effective contraception
* failure of acute or chronic severe organ
* hardly speak French and / or difficult to understand French

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a consultation with an allergist at the University Hospital of Nantes or city firm under a monitoring or an initial consultation for atopic dermatitis, allergic asthma or allergic rhinitis.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
average percentage of double positive T cells CD4 + / CD8 + compared to the average percentages of total T lymphocytes (CD3 +), CD4 + and the total number of peripheral blood formed elements | 3 months
  Intermediate biospecimen storage and preparation before centralized analyses

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Pays de la Loire Region, France

IPD SHARING:
Plan to Share IPD: Undecided